CLINICAL TRIAL: NCT06528522
Title: Impact of Smoking on Salivary Inflammatory Cytokines (Interleukin (IL)-39, IL-41, IL-1β, TNF-α) in Periodontal Disease
Brief Title: Impact of Smoking on Salivary Interleukin (IL)-39, IL-41, IL-1β, TNF-α Levels in Periodontal Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Osman Babayigit, Assistant Professor, Necmettin Erbakan University
Other Study IDs: IL-39-41-Smoke-Periodontitis
Record Dates: First submitted 2024-07-12; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis, Adult; Smoking; Periodontal Diseases
Keywords: periodontitis; cytokines; saliva
MeSH Terms: conditions — Chronic Periodontitis; Smoking; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-smoking - periodontally healthy: Participants eligible for inclusion are those who have reported a lifetime history of never smoking and exhibit periodontal health.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection
- smoking - periodontally healthy: Tobacco Use: Participants must have a documented history of smoking more than 10 cigarettes per day.
  Periodontal Health: Participants must exhibit clinically verified periodontal health, characterized by the absence of clinical attachment loss, probing depths within normal ranges, and no radiographic evidence of alveolar bone loss.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection
- non-smoking - periodontitis: Non-smokers: Only participants who have reported never smoking will be considered.
  Clinical Attachment Loss: Participants must exhibit a clinical attachment loss (CAL) of ≥3 mm in more than 30% of sites.
  Probing Depth: A probing depth (PD) of ≥5 mm must be present in at least six teeth.
  Radiographic Bone Loss: Participants must show radiographic evidence of bone loss extending to or beyond the middle third of the root in the coronal third.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection
- smoking - periodontitis: Smoking History: Participants must have reported smoking more than 10 cigarettes per day for a period exceeding 5 years.
  Clinical Attachment Loss (CAL): Participants must exhibit a clinical attachment loss of ≥3 mm in more than 30% of examined sites.
  Probing Depth (PD): A probing depth of ≥5 mm must be present in at least six teeth.
  Radiographic Bone Loss: Participants must demonstrate radiographic evidence of bone loss extending to or beyond the middle third of the root in the coronal third.
  Interventions: Diagnostic Test: Clinical Measurements and Saliva Sample Collection

INTERVENTIONS:
Diagnostic Test: Clinical Measurements and Saliva Sample Collection — Saliva samples will be collected from all participants, and comprehensive clinical parameters will be meticulously documented. The Plaque Index (PI) and Gingival Index (GI) will be measured at four sites per tooth. Full-mouth probing depth (PD) and clinical attachment level (CAL) will be recorded in detail for each tooth at six sites. The percentage of bleeding areas will be assessed within 20 seconds post-probing using a binary scoring system to indicate presence or absence. All clinical parameters will be recorded by a calibrated periodontologist utilizing manual probing techniques.
  Following collection, saliva samples will be stored at -80°C until subsequent analysis. Concentrations of IL-39, IL-41, IL-1β, and TNF-α in the saliva samples will be quantified using specific enzyme-linked immunosorbent assay (ELISA) kits.

SUMMARY:
The goal of this observational study is to evaluate if the measurement of salivary Interleukin (IL)-39, IL-41, IL-1Beta(β), and Tumor necrosis factor-alpha (TNF-α) levels can aid in the early diagnosis of periodontitis in patients with varying periodontal conditions, both smokers and non-smokers. The main questions it aims to answer are:

Can salivary IL-39, IL-41, IL-1β, and TNF-α levels be used as biomarkers for the early diagnosis of periodontitis? How do IL-41 and IL-39 levels correlate with smoking status in periodontal healthy and periodontitis patients? Researchers will compare the salivary biomarker levels between smokers and non-smokers to see if smoking affects these levels.

Participants will:

Provide salivary samples for biomarker analysis. Undergo a comprehensive periodontal examination to determine their periodontal status.

ELIGIBILITY:
Inclusion Criteria:

* The periodontitis groups (Non-smoking and smoking) in the study will include systemically healthy patients who are clinically diagnosed with Stage II and III, generalized, Grade B, C periodontitis based on the consensus report of the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions.
* Agreeing to participate in the study

Exclusion Criteria:

* use of oral contraceptive drugs
* use of antibiotics, immunosuppressants, or drug therapies in the last 6 months before the study;
* history of excessive alcohol use;
* pregnancy or breastfeeding status;
* periodontal treatment during the last 6 months before the study.
* Not agreeing to participate in the study
* Not meeting the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is planned to be conducted with 100 individuals aged between 18 and 65 who apply to the Department of Periodontology, Faculty of Dentistry, Necmettin Erbakan University, for various reasons. The eligibility of individuals to be included will be evaluated by Assistant Professor Dr. Osman BABAYIGIT at the Periodontology Clinic of NEU Faculty of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Periodontal clinical parameters (plaque index (PI)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include plaque index (PI) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Plaque Index (PI) Unit: Numerical score
Levels of IL-39, IL-41, IL-1β, and TNF-α saliva samples | baseline
  Levels of IL-39, IL-41, IL-1β, and TNF-α saliva samples (ng/L) Unit: Picograms per milliliter (pg/mL)
  IL-39, IL-41, IL-1β, and TNF-α levels will be assayed with commercially available kits using the enzyme-linked immunosorbent assay (ELISA) method.
Periodontal clinical parameters (percentage bleeding on probing (BOP)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include percentage bleeding on probing (BOP) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Percentage Bleeding on Probing (BOP) Unit: Percentage (%)
Periodontal clinical parameters (Clinical Attachment Level (CAL)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include clinical attachment level (CAL) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Clinical Attachment Level (CAL) Unit: Millimeters (mm)
Periodontal clinical parameters (gingival index (GI)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include gingival index (GI) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Gingival Index (GI) Unit: Numerical score
Periodontal clinical parameters (Probing Pocket Depth (PPD)) | baseline
  The measurements will be performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and will include probing pocket depth (PPD) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.
  Probing Pocket Depth (PPD) Unit: Millimeters (mm)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Babayigit O, Eroglu ZT, Sen DO, Sarac F, Altun S, Yarkac FU. Impact of smoking and periodontitis on salivary IL-39, IL-41, IL-1beta, and TNF-alpha levels: a cross-sectional analysis. BMC Oral Health. 2026 Jan 12. doi: 10.1186/s12903-026-07653-8. Online ahead of print. PMID 41527054